CLINICAL TRIAL: NCT01601717
Title: RTI-336 for Methamphetamine Dependence
Brief Title: RTI-336 as a Treatment for Methamphetamine Dependence
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Richard De La Garza, Associate Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: H-25186; 1R01DA027134 (NIH); DPMC (Other: NIDA)
Expanded Access: Available
Record Dates: First submitted 2009-12-10; First posted 2012-05-18 (Estimated); Last update posted 2012-05-18 (Estimated); Status verified 2012-05

CONDITIONS: Methamphetamine Dependence; Substance Abuse; Methamphetamine Abuse
Keywords: RTI-336; Methamphetamine
MeSH Terms: conditions — Substance-Related Disorders | interventions — 3beta-(4-chlorophenyl) tropane-2beta-(3-(4'-methylphenyl) isoxazol-5-yl) hydrochloride; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sugar pill (Placebo Comparator)
  Interventions: Drug: Placebo
- RTI-336 (Active Comparator)
  Interventions: Drug: RTI-336

INTERVENTIONS:
Drug: RTI-336 — Four medication dosage groups (0 mg, 1 mg, 12 mg, 20 mg) administered in the form of a pill once per day for 10 days.
  Arms: RTI-336
Drug: Placebo — Matching placebo pill administered once per day for 10 days.
  Other Names: Sugar pill
  Arms: Sugar pill

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of RTI-336 as a treatment for methamphetamine (METH) dependence in non-treatment-seeking METH-dependent volunteers.

DETAILED DESCRIPTION:
Methamphetamine (METH) is a highly addictive stimulant and acute exposure causes dopamine (DA) release and stimulates midbrain reward centers. The proposed work represents an important research effort with considerable public health significance in that it will evaluate a compound targeted specifically at DA transporter (DAT) inhibition for the treatment of METH dependence. The knowledge gained may ultimately support development and implementation of evidence-based treatments for METH dependence, a drug abuse problem with tremendous public health impact.

One therapeutic strategy is to develop and test compounds that normalize (increase) DA to determine if treatment with these drugs reduces METH use. A similar approach has been proposed as a treatment for cocaine dependence (Howell and Wilcox 2001; Mello and Negus 1996), another disorder associated with abnormally low DA activity (Martinez et al. 2007). In an effort to identify a DAT selective inhibitor, a number of 3-phenyltropane analogs were synthesized by RTI International. Among these, preclinical studies have shown that RTI-336 produced cocaine-like discriminative stimulus effects and reduced cocaine self-administration in rats, and produced dose-dependent suppression of cocaine self-administration in rhesus monkeys.

RTI-336 recently received IND-approval (75,778) for preliminary safety testing in healthy male volunteers, and is scheduled to be completed by February 2009. Subsequent to this effort, RTI-336 will be evaluated in a phase I trial involving cocaine-dependent volunteers. The current application puts forth, for the first time, a proposal to evaluate the preliminary efficacy of this very promising candidate medication in non-treatment-seeking METH-dependent volunteers.

ELIGIBILITY:
Inclusion Criteria:

In order to participate in the study, participants must:

1. Be English-speaking volunteers who are not seeking abstinence-focused treatment at the time of the study.
2. Be between 18-55 years of age.
3. Meet DSM-IV-TR criteria for METH dependence.
4. Self-report that preferred route of METH use is intravenous.
5. Have vital signs as follows: resting pulse between 50-90 bpm, blood pressure between 85-150 mmHg systolic and 45-90 mmHg diastolic.
6. Have a breathalyzer test indicating an undetectable blood alcohol level upon admission.
7. Have hematology and chemistry laboratory tests that are within normal ("b10%) limits with the following exceptions: Liver function tests (total bilirubin, ALT, AST, and alkaline phosphatase) < 3 x the upper limit of normal; Kidney function tests (creatinine and BUN) < 2 x the upper limit of normal
8. Have a baseline ECG that demonstrates normal sinus rhythm, normal conduction, and no clinically significant arrhythmias.
9. Have a medical history and brief physical examination demonstrating no clinically significant contraindications for study participation, in the judgment of the admitting physician and the principal investigator.
10. Weigh between 60 and 100 kg.

Exclusion Criteria:

Potential participants will be excluded from participation in the study if any of the following apply:

1. Have any previous medically adverse reaction to MA, including loss of consciousness, chest pain, or epileptic seizure.
2. Have neurological or psychiatric disorders, as assessed by MINI, such as: episode of major depression within the past 2 years; lifetime history of schizophrenia, other psychotic illness, or bipolar illness; current organic brain disease or dementia assessed by clinical interview; history of or any current psychiatric disorder which would require ongoing treatment or which would make study compliance difficult; history of suicide attempts within the past three months and/or current suicidal ideation/plan; history of psychosis occurring in the absence of current METH use.
3. Meet DSM-IV criteria for abuse/dependence on alcohol or other drugs, except nicotine or marijuana.
4. Have evidence of clinically significant heart disease or hypertension, as determined by physician.
5. Have evidence of untreated or unstable medical illness including: neuroendocrine, autoimmune, renal, hepatic, or active infectious disease.
6. Have HIV and currently symptomatic, have a diagnosis of AIDS, or currently taking antiretroviral medication.
7. Be pregnant or nursing. Other females must either be unable to conceive (i.e., surgically sterilized, sterile, or post-menopausal) or be using a reliable form of contraception (e.g., abstinence, birth control pills, intrauterine device, condoms, or spermicide). All females must provide negative pregnancy urine tests before study entry, and throughout the study.
8. Have any history of asthma, chronic coughing and wheezing, or other chronic respiratory illnesses.
9. Currently use alpha or beta agonists, theophylline, or other sympathomimetics.
10. Have any other illness, condition, or use of medications, which in the opinion of the PI and/or the admitting physician would preclude safe and/or successful completion of study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2010-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
The effects of RTI-336 and methamphetamine on cardiovascular measures
  Before and after each methamphetamine infusion during treatment with RTI-336, physiologic responses will be closely monitored using repeated HR, BP, and ECG readings. To evaluate safety, a DSMB will meet annually and following any serious AE to examine data as well as any new published information on RTI-336 relevant to the project. The number of AEs (including arrhythmias and ECG changes), changes in BP and HR, and changes in mood and psychiatric symptoms (using the BSI, BDI, POMS, and BPRS) will also be assessed throughout the study.

SECONDARY OUTCOMES:
The effects of RTI-336 and methamphetamine on subjective measures
  The ability of RTI-336 (1, 12 or 20 mg), as compared to placebo, to attenuate METH-induced (0 and 50 mg, IV) positive subjective effects (craving and ability to reduce reinforcing effects produced by methamphetamine) will be measured by: 1. VAS, Adjective Scales, and MCQ; 2. Choices for methamphetamine vs. money in the self-administration assay.

CONTACTS AND LOCATIONS:
Overall Officials: Richard De La Garza, PhD, Principal Investigator — Baylor College of Medicine